CLINICAL TRIAL: NCT07393841
Title: Molecular Indicators of Systematic Fitness
Acronym: MISFIT
Status: Recruiting | Type: Observational
Sponsor: VO Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 9554ed94-872a-4b5c-8a42-13e51f
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Adult; Fitness Testing; Athlete; Aging; Exercise Physiology; Human Performance
Keywords: VO2peak; VO2max; cardiorespiratory fitness; proteomics; blood biomarkers; cardiovascular health; oxygen transport; exercise performance; functional capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — The investigators are retaining two types of plasma (K2 EDTA and protease inhibitor tubes), serum, and whole blood (PAXgene).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention. — The investigators are not administering an intervention for this study. To opportunistically capture prospective data, the investigators give participants the option for re-testing after a period of time where participants are undergoing a self-directed intervention (i.e., no influence of the research staff), such as training for a marathon or other fitness event.

SUMMARY:
The goal of this study is to characterize associations between cardiorespiratory fitness, as measured by VO₂max/VO₂peak, and blood-based molecular measurements in adults. This is an observational study where research staff measures VO₂max/VO₂peak and collects fasted, resting blood samples on the same day. The main questions it aims to answer are:

1. Can a multi-analyte blood panel accurately predict directly measured VO₂max/VO₂peak?
2. How do these blood-based features vary across age, sex, and self-reported or documented physical activity profiles?
3. Are the predictor analytes able to capture changes in VO₂max/VO₂peak caused by a self-directed intervention (e.g., training for a marathon)?
4. What is the analytic reliability of the predictor biomarkers?

DETAILED DESCRIPTION:
Prospective observational cohort with baseline cross-sectional assessment; optional longitudinal follow-up with repeat VO₂max and blood collection in a subset. No intervention is assigned by the investigators. The investigators are amassing a large dataset of diverse individuals with directly measured VO2max paired with blood samples to support robust biomarker development.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥18 years old
* Be able to understand and provide informed consent (English; additional languages may be added via amendment with translated materials)
* Be willing to complete VO₂max testing, blood draw, and questionnaires.
* Be able to safely perform maximal/symptom-limited exercise testing as determined by: PAR-Q+ screening and investigator review (included as an attachment) and resting vitals screening (heart rate)

Exclusion Criteria:

* Conditions that, in the investigator's judgment, or a medical doctor, makes maximal exercise testing unsafe (e.g., unstable cardiovascular symptoms)
* Contraindications or unwillingness to undergo venipuncture
* Acute illness (fever, significant respiratory illness) at the time of testing
* Failure to comply with procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adults from the general community who are interested in health and fitness assessment. Participants are anticipated to primarily be athletes or recreational exercisers. This study does not specifically target clinical populations; however, individuals with stable medical conditions may participate if they have documented medical clearance to safely undergo maximal exercise testing.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2028-01-05 (Estimated); Study Completion 2028-05-10 (Estimated)

PRIMARY OUTCOMES:
A multi-analyte biomarker panel to predict maximal aerobic capacity | Day 1
  The primary outcome is developing a multi-protein biomarker panel that can accurately estimate cardiorespiratory fitness from the blood.
The change in VO2max/VO2peak and a multi-analyte biomarker panel after a self-directed training program. | From day 1 through study completion, average of 3 months
  In a subset of individuals who opt-in for a second study visit, the investigators will analyze the change in VO2max and the multi-analyte biomarker from pre- to post-testing.

CONTACTS AND LOCATIONS:
Locations (1):
- VO Health, Inc., New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared in order to protect participant privacy and confidentiality. The study was not designed with participant consent for public IPD sharing, and the data include sensitive physiological and molecular measurements. In addition, the collected data include proprietary measurements, algorithms, and analyses that are considered confidential and commercially sensitive. Only aggregate, de-identified results will be disseminated.